CLINICAL TRIAL: NCT01649362
Title: Effects of Prefeeding Oral Stimulation on Feeding Performance in Preterm Infants Born Between 26 and 33+6 Weeks' Gestational Age: a Case-control Study
Brief Title: Effects of Prefeeding Oral Stimulation on Feeding Performance in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier du Luxembourg (Other)
Collaborators: Luxembourg Institute of Health (Other Government)
Responsible Party: Principal Investigator, Dr Manon BACHE, Paediatrician, Centre Hospitalier du Luxembourg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201105/04
Record Dates: First submitted 2012-07-18; First posted 2012-07-25 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-02

CONDITIONS: Preterm Infant; Oral Feeding Performance
Keywords: preterm infant; feeding difficulties; prefeeding oral stimulation
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): No prefeeding oral stimulation
  Infants in the control group received neither oral stimulation nor a pacifier before or during gavage feeding.
- Oral stimulation, interventional group (Experimental): Infants in the interventional group received pre-feeding oral stimulation. The intervention started on infants born within 32 gestational weeks when the patients were stable and tube-fed, receiving more than 100 ml/kg/day of milk. On infants born after 32 weeks, the intervention started immediately after clinical stability was achieved.
  The pre-feeding oral stimulation program consisted of a 15-minute stimulation program delivered by one of the eight trained nurses or one trained member from the medical staff in accordance with the stimulation program proposed by Fucile, Gisel and Lau.
  The stimulation program was administered 15 to 30 minutes prior to tube feeding, once daily for at least 10 days. The program was stopped when the infants attained more than three oral feedings per day. The program was interrupted if the infants were medically unstable and/or had episodes of desaturation, apnoea and/or bradycardia during the intervention
  Interventions: Other: prefeeding oral stimulation program

INTERVENTIONS:
Other: prefeeding oral stimulation program — The intervention will start at 32 weeks PMA in a medically stable infant feed by gavage feeding for the infants born before 32 weeks' gestational age, and, as soon as clinical stability is acquired, for the infants born after 32 weeks.
  The prefeeding oral stimulation program consists of a 15-minute stimulation program, delivered by the nurse or the medical staff, according to the stimulation program proposed by Fucile, Gisel and Lau. The program is going to be administered once a day for 14 consecutive days (for infants born before 32 weeks' gestational age), 15 to 30 minutes before a tube feeding. In infants born after 32 weeks' gestational age, stimulation program is going to be stopped when the infant attains 3 complete oral feedings by day.
  Arms: Oral stimulation, interventional group

SUMMARY:
The objective of this study is to evaluate the efficacy of an oral stimulation program on the length of the transition period in preterm infants (primary outcome), the length of hospital stay and the breastfeeding rates at discharge (secondary outcomes).

DETAILED DESCRIPTION:
Oral feeding issues in preterm infants are a growing concern for neonatologists because the difficulties preterm infants show in transitioning from tube to independent oral feeding lead to delayed hospital discharge, maternal stress and rising financial burden.

Safety in infant oral feeding implies minimal risk of aspiration and requires the adequate coordination of sucking, swallowing and respiration.

Sucking and swallowing are present in early foetal life, but the coordination of sucking with swallowing and breathing is not thought to occur before 34 weeks post-menstrual age (PMA). Thus, preterm infants tend to suck, swallow and breathe in an alternate, rather than coordinated fashion.

Accelerated maturation of sucking reflex and earlier readiness for bottle-feeding is reported when preterm neonates were given non-nutritive sucking (NNS) opportunities during gavage feeding. Recent evidence suggests that the sensory consequences associated with the production of NNS have beneficial effects on oral feeding performance and the development of specific sucking skills.

At present, it is customary for infants who have stable cardiopulmonary status to be introduced to oral feeding around 33 to 34 weeks PMA. They usually take days or weeks in the transition period of combined gavage and oral feeding before reaching full oral feeding.

Recent studies suggest that an oral stimulation program associated to NNS applied to preterm infants for at least 10 days in the period of full gavage feeding can facilitate their oral feeding progress, improves breastfeeding rates among preterm infants and decreases the length of stay.

A meta-analysis found that NNS decreases significantly the length of hospital stay in preterm infants with an acceleration of the transition from tube to bottle feeds and better bottle feeding performance, without any negative outcomes reported.

Actually, in our neonatal intensive care unit, preterm infants don't receive any oral stimulation or a pacifier to develop NNS before oral feeding introduction and they show frequently, even for the infants born after 32 weeks' gestational age, difficulties in the transitioning from tube to independent oral feeding.

In a prospective randomized controlled clinical trial, prefeeding oral stimulation will be compared with the conventional approach for oral feeding initiation.

Considering a 15 days follow-up for each patient after the introduction of oral feeding, an expected rate of patients performing the full oral feeding after 15 days of 95% in the stimulated group and of 70% in the non stimulated group, the minimal sample size needed to observe a difference between the two groups would be 37 patients in each group with a power of 80% and an alpha level of 5%.

A total of 74 preterm infants are going to be included from the neonatal intensive care unit at the Children's Hospital of the Centre Hospitalier de Luxembourg, Luxembourg.

The investigators are going to include preterm infants from 26 to 33+6 weeks' gestational age, as determined by date of last menstruation and first-trimester ultrasound. Prior informed consent is going to be obtained from the parents/guardians of the newborns for their participation in the study.

Infants' randomization, into an experimental and a control group, is going to be done when they reach 32 weeks PMA for the infants born before 32 weeks, and at birth for the infants born after 32 weeks' gestational age. The process is done using sequential numbers, kept in sealed, opaque, non-translucid envelopes. Randomization is going to be stratified based on gestational age ranges (26-27+6, 28-29+6, 30-31+6, 32-33+6) to ensure a similar gestational age distribution in the two groups.

Infants in the interventional group are going to receive a prefeeding oral stimulation (group 1), the infants in the control group (group 2) are neither being stimulated nor will them be proposed a pacifier before or gavage feeding.

The intervention will start at 32 weeks PMA in a medically stable infant feed by gavage feeding for the infants born before 32 weeks' gestational age, and, as soon as clinical stability is acquired, for the infants born after 32 weeks.

The investigators defined as a complete oral feeding a minimal quantity of 5 millilitres that the preterm infant has to drink in less than 10 minutes by bottle or by breastfeeding. These 5 millilitres are the usual quantity that a preterm baby born at 34 weeks' gestational age is able to drink by himself at each meal.

The program is going to be interrupted if infants are medically unstable and/or have any episodes of oxygen desaturation, apnoea and/or bradycardia during the intervention.

Gavage feeding will begin when the preterm infant is clinically stable in terms of hemodynamics and has presented peristalsis according to criteria established by the caretaker staff. Oral diet progress depends on infant's tolerance and will be about 20 ml/kg/day.

The change from gavage to oral feeding is going to be initiated at 34 weeks PMA, after the beginning of oral stimulation program in group 1.

The gavage feeding will be stopped and the orogastric tube removed, when the infant attains an oral feeding volume of more than 120 ml/kg/day. A weight lost of 5 % is authorized after stopping gavage feeding.

Full oral diet is defined by an oral intake of milk > 150 ml/kg/day, by bottle or by breastfeeding, for 3 consecutive days.

The expected benefits of this study are a reduction in the length of stay in our neonatal unit in the stimulated group, due to the reduction in the length of the transition period in these preterm infants. A minimisation of the hospitalization cost and a reduction in the parental stress can by expected with an earlier hospital discharge.

An increase of the breastfeeding rates at discharge is expected. With the improved feeding performance in the stimulated group, the maternal stress concerning breastfeeding is reduced and the risk of failure is smaller. A better mother-child attachment can be expected with this study.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants from 26 to 33+6 weeks' gestational age, as determined by date of last menstruation and first-trimester ultrasound, hospitalized in our neonatal unit.

Exclusion Criteria:

* Congenital malformations (chromosomal disorders, malformations of head and face, neurological, cardiac, digestive or pulmonary malformations)
* Severe asphyxia (hypoxic-ischemic encephalopathy)
* Presence of third or fourth degree intracranial haemorrhage
* Severe periventricular leukomalacia
* Severe chronic lung disease
* Severe hospital infection during the study period
* Necrotising enterocolitis during the study period
* Feeding interruption for more than 10 days during the study period
* Death during the study period
* Transfer to another hospital before discharge.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Lise Lair, Study Chair — Luxembourg Institute of Health
Locations (1):
- Service de néonatologie, Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg

REFERENCES:
- [Background] Amaizu N, Shulman R, Schanler R, Lau C. Maturation of oral feeding skills in preterm infants. Acta Paediatr. 2008 Jan;97(1):61-7. doi: 10.1111/j.1651-2227.2007.00548.x. Epub 2007 Dec 3. PMID 18052999
- [Background] Arvedson J, Clark H, Lazarus C, Schooling T, Frymark T. Evidence-based systematic review: effects of oral motor interventions on feeding and swallowing in preterm infants. Am J Speech Lang Pathol. 2010 Nov;19(4):321-40. doi: 10.1044/1058-0360(2010/09-0067). Epub 2010 Jul 9. PMID 20622046
- [Background] Barlow SM, Finan DS, Lee J, Chu S. Synthetic orocutaneous stimulation entrains preterm infants with feeding difficulties to suck. J Perinatol. 2008 Aug;28(8):541-8. doi: 10.1038/jp.2008.57. Epub 2008 Jun 12. PMID 18548084
- [Background] Bingham PM, Ashikaga T, Abbasi S. Prospective study of non-nutritive sucking and feeding skills in premature infants. Arch Dis Child Fetal Neonatal Ed. 2010 May;95(3):F194-200. doi: 10.1136/adc.2009.164186. Epub 2009 Nov 29. PMID 19948525
- [Background] Boiron M, Da Nobrega L, Roux S, Henrot A, Saliba E. Effects of oral stimulation and oral support on non-nutritive sucking and feeding performance in preterm infants. Dev Med Child Neurol. 2007 Jun;49(6):439-44. doi: 10.1111/j.1469-8749.2007.00439.x. PMID 17518930
- [Background] Fucile S, Gisel E, Lau C. Oral stimulation accelerates the transition from tube to oral feeding in preterm infants. J Pediatr. 2002 Aug;141(2):230-6. doi: 10.1067/mpd.2002.125731. PMID 12183719
- [Background] Fucile S, Gisel EG, Lau C. Effect of an oral stimulation program on sucking skill maturation of preterm infants. Dev Med Child Neurol. 2005 Mar;47(3):158-62. doi: 10.1017/s0012162205000290. PMID 15739719
- [Background] Pickler RH, Reyna BA. Effects of non-nutritive sucking on nutritive sucking, breathing, and behavior during bottle feedings of preterm infants. Adv Neonatal Care. 2004 Aug;4(4):226-34. doi: 10.1016/j.adnc.2004.05.005. PMID 15368215
- [Background] Pimenta HP, Moreira ME, Rocha AD, Gomes SC Jr, Pinto LW, Lucena SL. Effects of non-nutritive sucking and oral stimulation on breastfeeding rates for preterm, low birth weight infants: a randomized clinical trial. J Pediatr (Rio J). 2008 Sep-Oct;84(5):423-7. doi: 10.2223/JPED.1839. English, Portuguese. PMID 18923786
- [Background] Pinelli J, Symington A. Non-nutritive sucking for promoting physiologic stability and nutrition in preterm infants. Cochrane Database Syst Rev. 2005 Oct 19;(4):CD001071. doi: 10.1002/14651858.CD001071.pub2. PMID 16235279
- [Background] Poore M, Zimmerman E, Barlow SM, Wang J, Gu F. Patterned orocutaneous therapy improves sucking and oral feeding in preterm infants. Acta Paediatr. 2008 Jul;97(7):920-7. doi: 10.1111/j.1651-2227.2008.00825.x. Epub 2008 May 7. PMID 18462468
- [Background] Rocha AD, Moreira ME, Pimenta HP, Ramos JR, Lucena SL. A randomized study of the efficacy of sensory-motor-oral stimulation and non-nutritive sucking in very low birthweight infant. Early Hum Dev. 2007 Jun;83(6):385-8. doi: 10.1016/j.earlhumdev.2006.08.003. Epub 2006 Sep 18. PMID 16979854
- [Background] Stumm S, Barlow SM, Estep M, Lee J, Cannon S, Carlson J, Finan D. Respiratory Distress Syndrome Degrades the Fine Structure of the Non-Nutritive Suck In Preterm Infants. J Neonatal Nurs. 2008;14(1):9-16. doi: 10.1016/j.jnn.2007.11.001. PMID 19122873
- [Background] Lau C. [Development of oral feeding skills in the preterm infant]. Arch Pediatr. 2007 Sep;14 Suppl 1:S35-41. doi: 10.1016/s0929-693x(07)80009-1. French. PMID 17939956

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: no prefeeding oral stimulation
- Oral Stimulation: preterm infants receiving an prefeeding oral stimulation program
Period: Overall Study
Arm/Group | Control Group | Oral Stimulation
Started | 47 | 54
Completed | 46 | 40
Not Completed | 1 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Oral Stimulation | Total
Number analyzed (Participants) | 46 | 40 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 46 | 40 | 86
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Customized [Mean (Standard Deviation); unit: weeks' gestational age] | 31.3 (1.7) | 31.4 (1.5) | 31.3 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 25 | 25 | 50
Region of Enrollment [Number; unit: participants]
  Luxembourg | 46 | 40 | 86

OUTCOME MEASURES:

1. Primary Outcome: Length of Transition Period
Description: transition period was defined as the period from the introduction of enteral feeding to full enteral feeding
Time Frame: participants were followed from date of randomization until full enteral feeding was acquired,an expected average of 5 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Group | Oral Stimulation
Number analyzed (Participants) | 46 | 40
days | 16.0 (6.9) | 16.9 (9.2)
Statistical Analysis 1: Comparison: Control Group vs Oral Stimulation; Test type: Superiority or Other; p = 0.63, t-test, 2 sided

2. Secondary Outcome: Length of Hospital Stay
Time Frame: participants were followed for the duration of hospital stay, an expected average of 5 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control Group | Oral Stimulation
Number analyzed (Participants) | 46 | 40
days | 42.5 (15.1) | 45.7 (16.8)
Statistical Analysis 1: Comparison: Control Group vs Oral Stimulation; Test type: Superiority or Other; p = 0.36, t-test, 2 sided

3. Secondary Outcome: Breastfeeding Rate at Discharge
Time Frame: hospital discharge, an expected average of 5 weeks from the beginning of oral feeding introduction
Measure: Number; unit: participants
Arm/Group | Control Group | Oral Stimulation
Number analyzed (Participants) | 46 | 40
participants | 21 | 28
Statistical Analysis 1: Comparison: Control Group vs Oral Stimulation; Test type: Superiority or Other; p = 0.02, Chi-squared

ADVERSE EVENTS:
Arm/Group | Control Group | Oral Stimulation
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/40
Other Adverse Events (participants affected / at risk) | 0/46 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No